CLINICAL TRIAL: NCT05274542
Title: Acute Effect of Blood Flow Restricted High-Intensity Resistive Training on Rectus Femoris Muscle Activity, Reaction Time, Muscular Performance, and Fatigue Level
Brief Title: Acute Effect of Blood Flow Restricted High-Intensity Resistive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Gülsena Utku, Principal Investigator, Halic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HI-BFR training
Record Dates: First submitted 2022-02-19; First posted 2022-03-10 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: High-Intensity Interval Training; Blood Flow Restriction Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity with blood flow restriction group (Experimental)
  Interventions: Other: high intensity with blood flow restriction
- high intensity without blood flow restriction group (Active Comparator)
  Interventions: Other: high intensity without blood flow restriction group

INTERVENTIONS:
Other: high intensity with blood flow restriction — Participants in high intensity with blood flow restriction group (n=12) will be given high-intensity resistance exercise training that restricts blood flow. Open kinetic chain rectus femoris resistance exercise training will be given with free weights, 80% of 1 RM with 8 repetitions, 2 sets and 3 minutes rest between sets. The exercises will be performed in a single session accompanied by a physiotherapist. A blood pressure cuff will be used to restrict blood flow. By applying the cuff to the proximal of the muscle, the blood flow will be restricted with a pressure of 150 mmHg and the muscle will be exercised in this way. After the exercise, the cuff will be removed and evaluations will be made after 2 minutes of rest.
  Arms: high intensity with blood flow restriction group
Other: high intensity without blood flow restriction group — Participants in high intensity without blood flow restriction group (n=12) will be given high-intensity resistance exercise training. Open kinetic chain rectus femoris resistance exercise training will be given with free weights, 80% of 1 RM with 8 repetitions, 2 sets and 3 minutes rest between sets. The exercises will be performed in a single session accompanied by a physiotherapist. After the exercise, after 2 minutes of rest, evaluations will be made.
  Arms: high intensity without blood flow restriction group

SUMMARY:
Recommended by many professional organizations such as the American College of Sports Medicine (ACSM) and the National Strength and Conditioning Association (NSCA), resistance exercise training improves muscle strength, body composition, performance, functionality and quality of life in healthy young adults. Blood flow restriction (BFR), also known as Kaatsu training, is proposed as a new method to improve muscle strength and muscle hypertrophy in a short time. Although there are studies in the literature in which BFR is applied with low-intensity resistance training, no studies have been found examining the effects of BFR applied with high-intensity resistance training on the neuromuscular adaptations of the quadriceps femoris muscle. Determining whether high-intensity resistance training with BFR is more effective on the quadriceps femoris muscle compared to high-intensity resistance training applied without BFR may provide faster and more effective responses by arranging resistance training protocols in terms of neuromuscular gains. Between 07.03.2022 and 07.06.2022, in the Biruni University Physiotherapy and Rehabilitation Department Application Laboratory, in which 24 healthy young adults between the ages of 18-25 (from 12 BFR, 12 BFR) will be included, exercise training to be applied with and without BFR was determined. Its effects will be compared with electromyographic measurement, single leg squat test, and measurement of late-onset muscle pain (Visual Analog Scale). IBM SPSS 21.0 statistical program will be used for statistical analysis. Whether the variables are suitable for normal distribution will be analyzed with the Shapiro-Wilk test. If the variables show normal distribution, the variation within the group will be analyzed with the paired samples t test, and if it does not show normal distribution, the Wilcoxon Signed rank test will be analyzed. Comparison of groups will be made with independent samples t-test in independent groups if the variables show normal distribution, and with Mann Whitney-U test if they do not show normal distribution. Categorical data distributions will be evaluated with the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25
* Healthy
* Be volunteer to participate the study

Exclusion Criteria:

* Pregnancy
* Breastfeeding status
* Cardiovascular disease
* Musculoskeletal problems
* Orthopedic problems related to the lower extremities
* Peripheral or central neurological disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
EMG measurement | immediately after intervention
  Electrodes in the RF muscle are placed in the middle of the muscle abdominals according to the recommendations of the Surface Electromyography for Non-Invasive Evaluation of Muscles club and the International Society of Electrophysiology and Kinesiology. Data will be evaluated with the Neurotrac® Simplex (Verity Medical Ltd., Braishfield, UK) wireless EMG device. The recording range in the device is between 0.2 µV - 2000 µV and has a 0.1 µV RMS sensitivity, 10 m free wireless (Bluetooth) connection range. The signals coming from the electrodes will be automatically filtered and transferred to digital media via software.

CONTACTS AND LOCATIONS:
Overall Officials: Gülsena Utku Umut, Principal Investigator — Halic University
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Derived] Korkmaz Dayican D, Ulker Eksi B, Yigit S, Utku Umut G, Ozyurek B, Yilmaz HE, Akinci B. Immediate Effects of High-Intensity Blood Flow Restriction Training on Muscle Performance and Muscle Soreness. Res Q Exerc Sport. 2025 Mar;96(1):213-222. doi: 10.1080/02701367.2024.2389902. Epub 2024 Aug 26. PMID 39186458
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/21922259/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/11018445/